CLINICAL TRIAL: NCT00582452
Title: Attitudes Towards Prophylactic Colectomy in HNPCC Patients
Brief Title: Attitudes Towards Prophylactic Colectomy in Hereditary Non-polyposis Colorectal Cancer (HNPCC) Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Karen Hurley, PhD, Memorial Sloan Kettering Cancer Center
Other Study IDs: 04-127; NCI CA101511; CA109236
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Cancer
Keywords: HNPCC; prophylactic colectomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 2: Affected patients who are at high risk for metachronous colorectal tumors due to mutation status.
  Interventions: Other: Telephone survey
- 1: Unaffected patients who are at high risk for developing colon cancer based on family history and/or mutation status.
  Interventions: Other: Telephone survey

INTERVENTIONS:
Other: Telephone survey — Telephone survey

SUMMARY:
The purpose of this study is to learn more about individual's with a family history of colon cancer and the process by which they may decide to undergo or not undergo prophylactic colectomy. This is a surgery to remove the colon in order to reduce risk of cancer (or of getting cancer again).

DETAILED DESCRIPTION:
Hereditary non-polyposis colorectal cancer (HNPCC) is associated with up to an 80% lifetime risk of developing colorectal cancer and a 40-50% chance of a metachronous tumor after partial colectomy for the disease. For these patients, prophylactic colectomy has been proposed as a potential risk management alternative to a lifetime of intensive surveillance by colonoscopy. The highly personal nature of such risk management decisions has been recognized in the development of individualized genetic counseling services. However, prior psychosocial research in this area has tended to use linear statistical techniques in which clinically important details are lost in an overly broad, one size-fits-all model that is difficult to apply in a one-to-one counseling session. We propose an innovative approach based on the Cognitive-Social Health Information Processing (C-SHIP) model in which we will explore how attitudes towards prophylactic colectomy are organized into meaningful patterns or types that can translate readily into tailored counseling recommendations. Specific aims of this study are: 1)to assess levels of intention in prophylactic colectomy among HNPCC patients; 2)To identify distinctive decision types based on profiles of perceived pros and cons of prophylactic colectomy; and 3) To explore the pattern of relations between decision types and counseling-related outcomes (level of intention in colectomy, cancer-specific anxiety, and colonoscopy adherence). We will conduct a one-time cross-sectional telephone survey of 320 HNPCC patients (defined as either carriers of a mutated mismatch repair gene associated with HNPCC or those with a personal/family history meeting published criteria for HNPCC). Using cluster analysis we will create a taxonomy of decision types. Prior research leads us to expect at least three types: Disengaged, Risk-Focused, and Ambivalent. We hypothesize that each type will have a different pattern of relations with the outcome variables (e.g., Risk-focused types will show higher level of intention regarding surgery, high anxiety, low avoidance, and high colonoscopy adherence, whereas Ambivalent types will show higher level of intention regarding surgery, high anxiety, high avoidance, and low colonoscopy adherence). Understanding these patterns will enhance the ability of physicians, genetic counselors, and other providers to help their patients make well informed, thoughtful decisions about the preventive strategy that will best protect their health, emotional well-being, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* are from a family that has a known mismatch repair mutation; or
* meet Amsterdam I or Amsterdam II criteria that spell out the family and personal cancer history characteristics associated with HNPCC
* are considered at sufficiently high risk by their CRC specialty physician that prophylactic colectomy may be presented as an option (excluding FAP).

Amsterdam I Criteria

1. At least three relatives with a colorectal cancer and the following criteria:

   * One should be a first degree relative of the other two
   * At least two successive generations should be affected
   * At least one colorectal cancer should be diagnosed before the age of 50
   * Familial Adenomatous Polyposis (FAP) should be excluded in the colorectal cancer case(s), if any

   Amsterdam II Criteria (also known as Revised Amsterdam Criteria
2. At least three relatives with an HNPCC-associated cancer (colorectal cancer, cancer of the endometrium, small bowel, ureter, or renal pelvis) *:

   * One should be a first degree relative of the other two
   * At least two successive generations should be affected
   * At least one relative should be diagnosed before age 50
   * FAP should be excluded in the colorectal cancer case(s), if any *NOTE: ovarian cancer will also be considered an HNPCCassociated cancer as per Lynch et al (NEJM 2003)

Exclusion Criteria:

* non-English speaking
* under the age of 18
* are unable to give meaningful informed consent due to physical, psychiatric or cognitive disability
* are from a family affected by FAP
* have already undergone subtotal colectomy or total proctocolectomy
* are in active treatment and/or less than six months post-surgery for cancer.
* Have undergone genetic counseling and testing for HNPCC at MSKCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unaffected patients who are at high risk for developing colon cancer based on family history and/or mutation status, and affected patients who are at high risk for metachronous colorectal tumors due to mutation status.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess levels of intention in prophylactic colectomy among individuals at increased familial risk of colorectal cancer and to identify distinctive decision types based on profiles of perceived pros and cons of prophylactic colectomy; | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hurley, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org